CLINICAL TRIAL: NCT03292341
Title: Evaluating a Decision Aid in Clinical Practice for Patients With T3/T4 Laryngeal Cancer
Brief Title: Evaluation of a Web-based Decision Aid Tool for Larynx Cancer (T3/T4) Patients.
Acronym: LaDecA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other); The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-28-03/06
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Larynx Cancer
MeSH Terms: conditions — Laryngeal Neoplasms | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients (Experimental): Patients diagnosed with larynx cancer and ex-larynx cancer patients:
  * Interviews with patients to define their decisional needs and to determine the barriers and facilitators to the implementation of shared decision making and the decision aid.
  * Navigating through the Treatmentchoice Decisional Tool and think aloud while running the tool
  * Questionnaires
  Interventions: Other: Interviews; Other: Treatmentchoice Decisional Tool; Other: Questionnaires
- Clinicians (Experimental): 2.Clinicians Radiotherapy-oncologists, ENT(Ear-Nose-Throat)-specialists, General practitioners, Nurses
  * Interviews with patients to define their decisional needs and to determine the barriers and facilitators to the implementation of shared decision making and the decision aid.
  * Navigating through the Treatmentchoice Decisional Tool and think aloud while running the tool
  * Questionnaires
  Interventions: Other: Interviews; Other: Treatmentchoice Decisional Tool; Other: Questionnaires
- Other involved organizations (Experimental): Patient Organizations and insurance companies Interviews with stakeholders (patients, clinicians, nurses, GP's, patient organizations, insurance companies) to determine the barriers and facilitators to the implementation of shared decision making and the decision aid
  Interventions: Other: Interviews with stakeholders

INTERVENTIONS:
Other: Interviews — Interviews with patients, physicians and general practitioners (GPs) to define patients' decisional needs
  Arms: Clinicians; Patients
Other: Treatmentchoice Decisional Tool — Patients and physicians navigate through Treatmentchoice Decisional Tool and think aloud while running the tool
  Arms: Clinicians; Patients
Other: Questionnaires — Patients and physicians fill out questionnaires on the usual care, Delphi study
  Arms: Clinicians; Patients
Other: Interviews with stakeholders — Interviews with stakeholders Interviews with stakeholders (patients, clinicians, nurses, GP's, patient organizations, insurance companies) to determine the barriers and facilitators to the implementation of shared decision making and the decision aid.
  Arms: Other involved organizations

SUMMARY:
Patients diagnosed with T3/T4 laryngeal cancer in general have several treatment options available, including total laryngectomy and/or (chemo-) radition. In order to help these patients in the decision making process, MAASTRO CLINIC designed and developed a web-based decision aid tool (Treatmentchoice). The aim of this study is twofold: user-testing Treatmentchoice using a systematically development process and establish the impact of Treatmentchoice on the decision making process.

The study covers 4 chronological activities: 1. assess decisional needs of patients and clinicians, 2. testing patients' and clinicians comprehensibility, acceptability and usability on the alpha-version of the tool, 3. establish the impact of Treatmentchoice on knowledge, decisional conflict and the shared decision making process, as well as the extent clinicians involve patients in decision making and 4. development of an implementation and dissemination plan for shared decision making which is based on the evaluation of barriers and facilitators for the use of patients decision aid tools in clinical practice.

A mixed method will be used. It comprises structured interviews combined with think aloud and questionnaires with stakeholders involved in the whole process (patients, medical doctors, nurses, general practitioners, patient organizations, and insurance companies).

DETAILED DESCRIPTION:
Laryngeal cancer is the second most common head and neck cancer. Each year about 700 people are diagnosed with larynxcarcinoma in the Netherlands (Van Dijk et.al. 2013).

For patients with laryngeal cancer, various treatment options are available, including surgery, radiotherapy, chemotherapy and endoscopic (laser) treatment. Each option has its own benefits and side effects. The optimal treatment for patients having stage 3 or 4 laryngeal cancer is not unambiguously proven. Different treatment options cause different side effects that may impact the patients' health-related quality of life. The treatment of choice depends on preferences and personal values. In these preference-sensitive choices it is important to involve the patient in the decision-making process. In this process both the practitioner and the patient exchange information and collaborate in the decision, the physician knows more technical information about the disease, the treatment options and the side effects, the patient knows how the treatment options correspond with his lifestyle, values and preferences (Frosch DL and Kaplan RM, 1999; O'Connor AM, et.al. 2003; O'Connor AM, et.al., 2004).

Patient Decision Aids (PDAs) are tools that can help patients to get involved in decision making by clarifying treatment options, outcomes, and personal values. In the development process of a decision aid it is mandatory to follow a systematic and iterative approach to: (a) understand patient's decisional needs; (b) create prototypical tools; (c) evaluate these prototypes with patients and clinicians, and (d) use these results to improve the tool.

Considering the International Patient Decision Aid Standards (http://ipdas.ohri.ca/), we designed an initial prototype, called Treatmentchoice (http://www.treatmentchoice.info). These standards recommend assessing patients and doctors views in decisional needs, use this information to develop an alpha version of the PDA and validate it again with patients and doctors to create a beta version.

The aim of this project is user-testing the initial prototype of the Treatmentchoice. This will allow us to follow a systematically development process and to gain knowledge on the validity of our approach. The project covers 4 chronological activities:

ACTIVITY 1: ASSES DECISIONAL NEEDS: Elicit patients and clinicians views on patient's information, expectations, and needs on decision support. Conclusions and recommendations for improvement of Treatmentchoice will be derived and the current prototype will be improved creating an alpha prototype.

ACTIVITY 2: ALPHA-TESTING: Testing patients' and clinicians comprehensibility, acceptability and usability on the alpha-version. A mixed method will be used; structured interviews combined with think aloud (Ahmed, 2009) and questionnaires (Unified Theory of Acceptance and Use of Technology (UTAUT) - Venkatesh et al.2012) with both patients and clinicians (head and neck surgeon,medical oncologists an radiation oncologists). Conclusions and recommendations will be documented. Considering this assessment, the prototype will be improved. Alpha testing will be repeated with this improved prototype using an iterative process, until the tool is comprehensible, acceptable and usable for both patients and physicians. A second assessment will be performed with a beta prototype.

ACTIVITY 3: BETA-TESTING: Establish the impact of Treatmentchoice on knowledge, decisional conflict and the shared decision making process, as well as the extent clinicians involve patients in decision making. The study composes the evaluation of the impact of the Treatmentchoice. A variety of questionnaires will be used to assess different outcome measures:

* Age and educational level, home situation with regard to internet connection.
* Knowledge test will be assessed using 20 statements, which can be rated as "true", "not true" or "do not know" (Savelberg, 2015).
* Decisional conflict will be assessed using the Decisional Conflict Scale (DCS). This 16-item scale has five subscales: feeling informed, decisional uncertainty, clear values, support, and quality of decisions. Each of these items is scored on a five-point Likert scale from 1 (strongly agree) to 5 (strongly disagree) (DCS, O'Connor AM, 2010).
* Patient's desire to participate in medical decisions will be assessed using a 5-item Control Preference Scale (Degner 1997).
* The Shared Decision Making (SDM) process will be assessed by the perceptions of patients, using the SDM-Q9 instrument for patients. The instrument provides 9 statements, which can be rated on a six-point scale from 0 (completely disagree) to 5 (completely agree). (SDM-Q9, Rodenburg, 2015 Dutch version).
* The process of SDM will also be assessed by the perceptions of the physician (the oncologist or the radiotherapist if the decision is made together with the radiotherapist), using the SDM-Q9 instrument for professionals. The instrument provides 9 statements, also rated on a six-point scale (SDM-Q9,Rodenburg,2015/Dutch version).

The patients will be asked to fill in the questionnaires at two time points, directly after the decision making process and 3 months after the decision making process. Their physician will be asked to fill in the questionnaire at 1 time point, directly after the decision making process.

ACTIVITY 4: IMPLEMENTATION: Develop an implementation and dissemination plan for shared decision making in prostate cancer. Questionnaires and qualitative interviews will be performed to evaluate barriers and facilitators for implementation in clinical practice, to develop strategies for the implementation of the decision aid and facilitate optimal shared decision making, tailored to the barriers and needs of the end-users. Based on the results, an implementation plan will be written

ELIGIBILITY:
1. Larynx cancer patients

   Inclusion Criteria:
   * Larynx cancer: T3 anyN M0, T4 anyN M0
   * Proficient in Dutch
   * minimal 18 years old

   Exclusion Criteria:
   * Patients that do not have a treatment choice (due to contra-indications or other medical reasons)
   * patients with recurrent disease

   For alpha testing patients that already made there decision are selected. For each treatment option (external beam RT, surgery and chemoradiation) at least 10 patients will be included. For beta testing patients that are facing their decision will be included. Aiming for an effect size of 0.60 for a difference in mean total score on the Decisional Conflict Scale, it would require 45 patients per hospital (pre and post intervention) to determine this effect with alpha 0.05 and power 0.80.
2. Physicians

   * Radiotherapy-oncologists
   * Oncologists
   * General practitioners
   * Nurses For alpha testing at least 10 physicians are selected. For beta testing at least 45 questionnaires are required.
3. Patient organizations and insurance companies Besides patients and physicians, patient organizations and insurance companies will be involved to evaluate barriers and facilitators for implementation in clinical practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Patient's decisional needs to make a decision about their treatment | up to 1 year
  Patients' decisional needs (development phase):semi-structured interviews with patients about their medical history, their experience with the treatment, the decision about their treatment, and what information the patients need to make
Comprehensibility of the decision aid too | up to 1 year
  Quantitative research using the Unified Theory of Acceptance and Use of Technology (UTAUT Venkatesh et al. 2013). This questionnaire. (5-Likert) measure how patients and clinicians perceived its utility, effectiveness and efficiency for shared decision-making, as well as their satisfaction with the decision aid.
Usability of the decision aid too | up to 1 year
  Quantitative research using a questionnaire based on the International Standard ISO-9242-11. This questionnaire (5-Likert) measure to what extent the decision aid is easy to use.
Decisional conflict (patients, evaluation phase) | 2 weeks after diagnosis
  Decisional conflict will be assessed using the DCS (Decisional conflict scale): change in DCS between baseline group (usual care) and intervention group (use of the aid tool)
Control Preference Scale (patients; evaluation phase) | 2 weeks after diagnosis
  Patient's preference to participate in medical decisions will be assessed using the 5-item Control Preference Scale (CPS):change in CPS between baseline group (usual care) and intervention group (use of the aid tool)
Perception shared decision-making (patients; evaluation phase) | 2 weeks after diagnosis
  Patient's perception of the shared decision-making process will be assessed using the (shared decision making) SDM-Q9 instrument for patients: change in SDM between baseline group (usual care) and the intervention group (use of the aid tool)
. Perception shared decision-making (doctors; evaluation phase) | 2 weeks after diagnosis
  Doctor's perception of the shared decision-making process will be assessed using the SDM-Q9 instrument for professionals: change in SDM between baseline group (usual care) and the intervention group (use of the aid tool)]]

SECONDARY OUTCOMES:
Patients' views on the current decision-making process | upto 1 year
  Patients' views on the current decision-making process (development phase)
Patients' satisfaction with decision aid (Treatmentchoice) | upto 1 year
  Patients' satisfaction with decision aid (Treatmentchoice) (development phase)
Patients' intention to use and recommend Treatmentchoice to others | an average of 2 year
  Patients' intention to use and recommend Treatmentchoice to others (development phase)
Insights into the value clarification process of prostate cancer patients | an average of 2 year
  Insights into the value clarification process of prostate cancer patients by questionnaires (development phase)

OTHER OUTCOMES:
Barriers and facilitators for the implementation of Treatmentchoice in clinical practice | an average of 2 years
  Barriers and facilitators for the implementation of Treatmentchoice in clinical practice (implementation phase) will be assessed by questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Frank Hoebers, MD,PhD, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- MAASTRO Clinic, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heirman AN, Petersen JF, Al-Mamgani A, Eerenstein SEJ, de Kleijn BJ, Hoebers F, Tijink BM, van der Molen L, Halmos GB, Dirven R, Stuiver MM, van den Brekel MWM. The impact of a patient decision aid for patients with advanced laryngeal carcinoma - a multicenter study. BMC Med Inform Decis Mak. 2025 Jul 1;25(1):217. doi: 10.1186/s12911-025-03080-x. PMID 40597116
- [Derived] Petersen JF, Berlanga A, Stuiver MM, Hamming-Vrieze O, Hoebers F, Lambin P, van den Brekel MWM. Improving decision making in larynx cancer by developing a decision aid: A mixed methods approach. Laryngoscope. 2019 Dec;129(12):2733-2739. doi: 10.1002/lary.27800. Epub 2019 Jan 21. PMID 30663068